CLINICAL TRIAL: NCT06516692
Title: (IVCIN TRIAL) Outcomes of Patient Admitted to Critical Care Unit with Vs Without Inferior Vena Cava Collapsibility and Distensibility Assessment. a Randomized Clinical Trial in Pakistan.
Brief Title: Inferior Vena Cava Collapsibility and Distensibility Assessment in Critical Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NO.F.2-81/2023-GENL/64/JPMC
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Sepsis; Acute Renal Failure; Acute Gastroenteritis; Diabetic Ketoacidosis
Keywords: Inferior Vena Cava Collapsibility and Distensibility index; Fluid management; Resuscitation; Clinical parameters; Sepsis; Acute gastroenteritis; Acute Renal failure; Diabetic ketoacidosis; Mortality; Cumulative fluid balance; Lactic acid; Sequential Organ Failure Assessment score; Mechanical Ventilation; Critical Care
MeSH Terms: conditions — Sepsis; Acute Kidney Injury; Diabetic Ketoacidosis | interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Clinical Parameters guided assessment arm (No Intervention): Participants recruited to this arm will be assessed for their hydration status and further fluid management as per usual care of assessment through
  * Capillary refill time
  * Presence/absence of pulmonary rales.
  * Jugular venous pressure assessment by clinical methods
  * Presence / absence of pedal edema
- Inferior Vena Cava Collapsibility and Distensibility guided assessment arm (Experimental): Participants recruited in this arm will be assessed through measurement of inferior vena cava diameter via subcostal window within 3 cm of its opening to right atrium through point of care ultrasound using a curvilinear or phased array probe.
  For spontaneously breathing patients Inferior Vena Cava Collapsibility Index (IVC CI) will be calculated as:
  [(IVC diameter max-IVC diameter min)/IVC diameter max]×100%
  * IVC CI > 50% = overt hypovolemia
  * IVC CI < 20% = no overt hypovolemia
  * IVC CI of 20% to 50% will be goal
  For mechanically ventilated patients Inferior Vena Cava Distensibility Index (IVC DI) will be calculated as:
  [(IVC diameter max-IVC diameter min)/IVC diameter min]×100% IVC distensibility>18% = hypovolemia IVC distensibility<18% = no hypovolemia
  Interventions: Diagnostic Test: Inferior Vena Cava Collapsibility/distensibility Index (IVC CI/DI) assessment

INTERVENTIONS:
Diagnostic Test: Inferior Vena Cava Collapsibility/distensibility Index (IVC CI/DI) assessment — Assessment of hydration status in critically ill patient recruited to this arm will be intervened through an ultrasound guided calculation of collapsibility and distensibility index of Inferior Vena Cava. This method of intervention will be continued and repeated as needed throughout the stay of the participant in intensive care unit.
  Arms: Inferior Vena Cava Collapsibility and Distensibility guided assessment arm

SUMMARY:
This study will help in determining the impact of assessment of Inferior Vena Cava Collapsibility and Distensibility Index (IVC CI and DI) through Point Of Care Ultra Sound (POCUS), for the fluid management of critically ill patients. This would help in better management of such patients in resource limited countries, where costly equipment for cardiac output monitoring and fluid management are frequently not available.

Moreover this study will help in development of future guidelines for fluid resuscitation in critically ill patients.

DETAILED DESCRIPTION:
The current study is a randomized clinical trial with the aim to explore comparative outcome between IVC CI and DI versus clinical parameters guided fluid management groups in patients of sepsis, Acute renal failure, Acute gastroenteritis and Diabetic ketoacidosis in terms of,

1. Within 24 hours 7 day and 28 day mortality
2. Change in Sequential Organ failure Assessment (ΔSOFA) score from baseline to 24 hours after fluid management.
3. Cumulative fluid balance at 6 hours of fluid management
4. Days on mechanical ventilation
5. Days in Intensive Care Unit (ICU)
6. Change in lactic acid levels in sepsis sub group
7. Change in Blood sugar Random (BSR) in Diabetic ketoacidosis (DKA) sub group
8. Change in Power of Hydrogen (PH) in septic and diabetic ketoacidosis sub group of participant

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in critical care with systolic Blood Pressure < 90 mmHg with any of the diagnosis as per operational definition:
* Sepsis
* Diabetic ketoacidosis
* Acute kidney injury
* Acute gastroenteritis

Exclusion Criteria:

* Known case of right heart disease
* Known case of congestive cardiac failure
* Presence of marked ascites
* IVC could not be identified or diameter could not be measured
* Pregnant females
* Body Mass Index (BMI) >30 Kg/meter2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Within 24-hours, 7-day and 28 day mortalities | Mortalities will be assessed and recorded within 24hour, then day 7 up to 28th day.
  Death of participant will be considered mortality.
Cumulative fluid balance | At 6 hours of enrolment of participant
  A difference of total amount of fluids given both intravenously and through oral rout to a total amount of urine output or fluid removed during dialysis, calculated in milliliter (ml) will be taken as cumulative fluid balance.
Change in Sequential Organ Failure Assessment score(Δ SOFA) | At 24 hours of enrolment
  A difference will be noted in initial Sequential Organ Failure Assessment score ( from 0 up to 24) to score at 24 hours .A positive difference in score will be considered as improvement and a negative difference will be considered as worsening in outcomes. Values for cumulative SOFA scores as well as individual organ SOFA scores for hepatic, neurological, cardiovascular, renal, coagulopathy and respiratory will be analyzed.

SECONDARY OUTCOMES:
Days in Intensive Care Unit (ICU) | ICU days up to 28 day
  Total ICU stay in days will be noted
Days on mechanical ventilation | Days in which participant will be on mechanical ventilation up to 28 days
  This outcome will be measured for the participants who will be mechanically ventilated.
Change in lactic acid levels in septic patient | At 6 hours of enrolment of participant
  This outcome will be measured as difference of values from the time of enrolment to 6 hours in mmol/L in patients with diagnosis of sepsis in the trial
Change in Blood Sugar random (BSR) levels in patients with diabetic ketoacidosis | At 6 hours of enrolment of participant
  This outcome will be measured in mg/dL in patients with diagnosis of diabetic ketoacidosis in the trial
Change in Power of hydrogen (PH) in patients with sepsis and diabetic ketoacidosis | At 6 hours of enrolment of participant
  This outcome will be calculated as difference of values from time of enrolment to 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Shamim Kausar, EDIC,FCPS, Principal Investigator — Jinnah Post Graduate and Medical Centre
Locations (1):
- Jinnah Post graduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan to share Individual patient data.

REFERENCES:
- [Background] Kashani K, Omer T, Shaw AD. The Intensivist's Perspective of Shock, Volume Management, and Hemodynamic Monitoring. Clin J Am Soc Nephrol. 2022 May;17(5):706-716. doi: 10.2215/CJN.14191021. Epub 2022 Apr 4. PMID 35379765
- [Background] Basmaji J, Arntfield R, Desai K, Lau VI, Lewis K, Rochwerg B, Fiorini K, Honarmand K, Slessarev M, Leligdowicz A, Park B, Prager R, Wong MYS, Jones PM, Ball IM, Orozco N, Meade M, Thabane L, Guyatt G. The Impact of Point-of-Care Ultrasound-Guided Resuscitation on Clinical Outcomes in Patients With Shock: A Systematic Review and Meta-Analysis. Crit Care Med. 2024 Nov 1;52(11):1661-1673. doi: 10.1097/CCM.0000000000006399. Epub 2024 Sep 18. PMID 39298556
- [Background] Musikatavorn K, Plitawanon P, Lumlertgul S, Narajeenron K, Rojanasarntikul D, Tarapan T, Saoraya J. Randomized Controlled Trial of Ultrasound-guided Fluid Resuscitation of Sepsis-Induced Hypoperfusion and Septic Shock. West J Emerg Med. 2021 Feb 10;22(2):369-378. doi: 10.5811/westjem.2020.11.48571. PMID 33856325
- [Background] Spiliotaki E, Saranteas T, Moschovaki N, Panagouli K, Pistioli E, Kitsinelis V, Briasoulis P, Papadimos T. Inferior vena cava ultrasonography in the assessment of intravascular volume status and fluid responsiveness in the emergency department and intensive care unit: A critical analysis review. J Clin Ultrasound. 2022 Jun;50(5):733-744. doi: 10.1002/jcu.23194. Epub 2022 Mar 18. PMID 35302241
- [Background] Kaptein EM, Kaptein MJ. Inferior vena cava ultrasound and other techniques for assessment of intravascular and extravascular volume: an update. Clin Kidney J. 2023 Jun 29;16(11):1861-1877. doi: 10.1093/ckj/sfad156. eCollection 2023 Nov. PMID 37915939
- See also: The Intensivist's Perspective of Shock, Volume Management, and Hemodynamic Monitoring — https://pubmed.ncbi.nlm.nih.gov/35379765/